CLINICAL TRIAL: NCT02208453
Title: A Single Arm, Open-label, Prospective, Study to Assess the Feasibility, Efficacy and Safety of InSpace™ Device Implantation in a Procedure Under Local Anesthesia for a Treatment of Subjects With Massive, Irreparable Rotator Cuff Tear
Brief Title: InSpace™ System Implantation in a Procedure Under Local Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OrthoSpace Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IS-CL-05; 72746 (Other: Santa Maria Della Miserecordia, Udine)
Record Dates: First submitted 2013-06-29; First posted 2014-08-05 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Rotator Cuff Tear
Keywords: Massive Rotator Cuff Tear; Local anesthesia; Sub-acromial spacer
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No

ARMS (1):
- InSpace implantation (Experimental): InSpace device implantation
  Interventions: Device: InSpace Implantation

INTERVENTIONS:
Device: InSpace Implantation — InSpace device Implantation

SUMMARY:
The study objective is to assess the feasibility, efficacy and safety of the InSpace™ Device implantation in a surgical procedure under local anesthesia using arthroscopic and/or fluoroscopic visualization of the affected shoulder.

DETAILED DESCRIPTION:
A single arm, open-label, prospective, study to assess the feasibility, efficacy and safety of InSpace™ device implantation in a procedure under local anesthesia for a treatment of subjects with massive, irreparable rotator cuff tear.

Subjects with radiological confirmed massive RCT who are eligible per inclusion/exclusion criteria, will be enrolled for the study treatment.

Subjects will undergo surgical intervention under local anesthesia , fluoroscopic and/ or arthroscopic visualization of InSpace™ implantation.

Subjects will then be followed for safety and efficacy for a 24 months following the implantation.

The study objective is to assess the feasibility, efficacy and safety of the InSpace™ Device implantation in a surgical procedure under local anesthesia using arthroscopic and/or fluoroscopic visualization of the affected shoulder.

The efficacy will be assess by using Constant and ASES outcome score The Constant and the ASES will be completed by the investigator at each study visit .The patient will complete the patient self-evaluation part of the ASES at each study visit.

The Safety assessment will be conducted by collecting all device related AEs/SAEs throughout the entire study period.

ELIGIBILITY:
Inclusion Criteria:

1. Age 50 or older.
2. Positive diagnostic MRI of the affected shoulder indicating full thickness massive irreparable RCT of at least 5cm in diameter (according to Cofield classification) including fatty infiltration grade III or IV (according to classification of Goutallier).
3. Persistent pain and failure of non-operative treatment of the affected shoulder for at least 3 months.

Exclusion Criteria:

1. Known allergy to the balloon material
2. Evidence of significant osteoarthritis or cartilage damage in the shoulder
3. Evidence of gleno-humeral instability
4. Evidence of major joint trauma, infection, or necrosis in the shoulder
5. Major medical condition or known drug or alcohol abuses that could affect quality of life and influence the results of the study.
6. Concurrent participation in any other invasive clinical study one month prior to enrollment to the study and during the entire study period.
7. Subjects with worker's compensation claims or other litigation claims related to the shoulder being treated in the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Change in total shoulder outcome scores (Constant and ASES) | 6 months post implanatation
  Change in total shoulder outcome scores (Constant and ASES)at 6 month post implantattion

SECONDARY OUTCOMES:
Change in Total Shoulder scores | up to 24 months post implantation
  Change in Total Shoulder scores and improvement compare to baseline at each time point (6W, 3m, 12m and 24m).

OTHER OUTCOMES:
Safety Assessment | 24 months post implantation
  The Safety assessment will include all device related AEs/SAEs throughout the entire study period.

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Gervasi, MD, Principal Investigator — Orthopedic Department, Latisana Hospital
Locations (1):
- Hospital of Latisana, Latisana, Udine, Italy

REFERENCES:
- See also: Fluoroscopy-guided biodegradable spacer implantation using local anesthesia: safety and efficacy study in patients with massive rotator cuff tears. — http://www.ncbi.nlm.nih.gov/pubmed/27900707